CLINICAL TRIAL: NCT00006240
Title: A Pilot Study of Phenylbutyrate, Dexamethasone and GM-CSF in Refractory or Relapsed t(8;21) Acute Myeloid Leukemia
Brief Title: Phenylbutyrate, Dexamethasone, and Sargramostim in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068165; NHLBI-00-H-0156; NCI-171
Record Dates: First submitted 2000-09-11; First posted 2003-07-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2002-11

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — sargramostim; Dexamethasone; 4-phenylbutyric acid

INTERVENTIONS:
Biological: sargramostim
Drug: dexamethasone
Drug: oral sodium phenylbutyrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combining phenylbutyrate, dexamethasone, and sargramostim in treating patients who have refractory or relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response (complete hematologic remission induction) of phenylbutyrate, dexamethasone, and sargramostim (GM-CSF) in patients with refractory or relapsed t(8;21) acute myeloid leukemia.
* Determine the correlation between histone acetylation, differentiation, and apoptosis in bone marrow mononuclear cells with response rate in patients treated with this regimen.
* Determine the overall survival of patients on this regimen.
* Determine the correlation between histone acetylation, differentiation, and apoptosis in bone marrow mononuclear cells with pharmacokinetics of this regimen in these patients.
* Determine the safety and toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive phenylbutyrate IV continuously and sargramostim (GM-CSF) subcutaneously on days 1-7 and 15-21. Patients also receive oral dexamethasone on days 1-4 and 15-18. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity until complete hematologic remission is induced. Patients with stable disease at the end of 1 course receive at least 2 additional courses.

Patients are followed twice a week for 3 months, monthly for 1 year, every three months for the next 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 9-24 patients will be accrued for this study in at least 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of t(8;21) acute myeloid leukemia (AML)

  * Failed standard induction chemotherapy or stem cell transplantation (SCT) OR
  * Relapsed after standard induction chemotherapy or SCT OR
  * Refused or not a candidate for SCT or matched allogeneic sibling bone marrow transplantation or donor lymphocyte infusion OR
  * Refused of not a candidate for autologous SCT or bone marrow transplantation
* No CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 7 days

Hematopoietic:

* Not specified

Hepatic:

* AST or ALT no greater than 3 times upper limit of normal (ULN)
* Bilirubin no greater than 3 times ULN
* No hepatic disease that would preclude study

Renal:

* Creatinine no greater than 2 mg/dL
* Creatinine clearance at least 60 mL/min
* No renal disease that would preclude study

Cardiovascular:

* No cardiac disease that would preclude study
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within past 8 weeks

Other:

* No active infection except cystitis
* Not pregnant or nursing
* No altered mental status or seizure disorder
* No other serious disease that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 3 weeks since prior investigational antineoplastic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Liu, MD, Study Chair — National Heart, Lung, and Blood Institute (NHLBI)
Locations (4):
- United States (4):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - National Heart, Lung, and Blood Institute, Bethesda, Maryland
  - Mount Sinai Medical Center, NY, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania